CLINICAL TRIAL: NCT06065540
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) s.c. in Doses 2.4/2.4 mg and 1.0/1.0 mg Once Weekly Versus Semaglutide 2.4 mg and 1.0 mg, Cagrilintide 2.4 mg and Placebo in Participants With Type 2 Diabetes Inadequately Controlled on Metformin With or Without an SGLT2 Inhibitor
Brief Title: A Research Study to See How Well CagriSema Compared to Semaglutide, Cagrilintide and Placebo Lowers Blood Sugar and Body Weight in People With Type 2 Diabetes Treated With Metformin With or Without an SGLT2 Inhibitor
Acronym: REIMAGINE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-4896; U1111-1283-0427 (Other: World Health Organization (WHO)); 2022-502678-18 (EudraCT Number)
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- CagriSema Dose 1 (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of cagrilintide dose 1 and semaglutide dose 1 for 68 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- CagriSema Dose 2 (Experimental): Participants will receive once-weekly s.c injections of cagrilintide dose 2 and semaglutide dose 2 for 68 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Semaglutide Dose 1 (Active Comparator): Participants will receive once-weekly s.c injection of semaglutide dose 1 for 68 weeks.
  Interventions: Drug: Semaglutide
- Semaglutide Dose 2 (Active Comparator): Participants will receive once-weekly s.c injection of semaglutide dose 2 for 68 weeks.
  Interventions: Drug: Semaglutide
- Cagrilintide Dose 1 (Active Comparator): Participants will receive once-weekly s.c injection of cagrilintide dose 1 for 68 weeks.
  Interventions: Drug: Cagrilintide
- Placebo Dose 1 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrilintide dose 1 and semaglutide dose 1 for 68 weeks.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide
- Placebo Dose 2 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrilintide dose 2 and semaglutide dose 2 for 68 weeks.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly s.c injection of cagrilintide at escalating doses every week until maintenance dose 1 and dose 2 of cagrilintide is reached.
  Arms: CagriSema Dose 1; CagriSema Dose 2; Cagrilintide Dose 1
Drug: Semaglutide — Participants will receive once-weekly s.c injection of semaglutide at escalating doses every week until maintenance dose 1 and dose 2 of semaglutide is reached.
  Arms: CagriSema Dose 1; CagriSema Dose 2; Semaglutide Dose 1; Semaglutide Dose 2
Drug: Placebo cagrilintide — Participants will receive placebo matched to cagrilintide subcutaneously.
  Arms: Placebo Dose 1; Placebo Dose 2
Drug: Placebo semaglutide — Participants will receive placebo matched to semaglutide subcutaneously.
  Arms: Placebo Dose 1; Placebo Dose 2

SUMMARY:
The study will look at how well CagriSema helps people lower their blood sugar and body weight. CagriSema is a new weekly medicine that combines two medicines called semaglutide and cagrilintide. CagriSema will be compared to the two medicines semaglutide and cagrilintide, when they are taken alone. CagriSema will also be compared to a "dummy" medicine without any active ingredient. The study will be done in participants who have type 2 diabetes. Participants will take the study medicine together with the current diabetes medicine (metformin with or without an SGLT2 inhibitor).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days before screening.
* Stable daily dose(s) greater than or equal to 90 days before screening of any of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator: metformin with or without Sodium-Glucose Cotransporter-2 (SGLT2) inhibitors.
* Glycated haemoglobin (HbA1c) 7.0-10.5 percent (53-91 millimoles per mole [mmol/mol]) (both inclusive) as determined by central laboratory at screening.
* Body Mass Index (BMI) greater than or equal to 25 kilogram per square metre ( kg/m^2) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening.

Exclusion Criteria:

* Renal impairment with estimated Glomerular Filtration Rate (eGFR) less than 30 milliliters per minute per 1.73 square metre (mL/min/1.73 m^2) as determined by central laboratory at screening.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2734 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
CagriSema (dose 1) versus semaglutide (dose 1): Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.

SECONDARY OUTCOMES:
CagriSema versus cagrilintide: Change in HbA1c | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus cagrilintide: Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage.
CagriSema (dose 1) versus semaglutide (dose 2): Change in HbA1c | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage.
Cagrilintide versus placebo: Change in HbA1c | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.
Cagrilintide versus placebo: Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage.
CagriSema versus semaglutide: Achievement of greater than or equal to (>=) 10 percent (%) weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants.
CagriSema versus semaglutide: Achievement of >= 15 % weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants.
CagriSema versus semaglutide: Achievement of >= 20 % weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants.
CagriSema (pooled doses) versus semaglutide (pooled doses): Continuous Glucose Monitoring (CGM) - Change in Time in Range (TIR) 3.9-10.0 millimoles per litre (mmol/L) (70-180 milligrams per decilitre [mg/dL]) | From baseline (week -3) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: CGM - Change in time in Tight Target Range (TITR) 3.9-7.8 (mmol/L) (70-140 mg/dL) | From baseline (week -3) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeters of mercury (mmHg).
CagriSema versus semaglutide: Ratio to baseline in triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of triglycerides.
CagriSema versus semaglutide: Ratio to baseline in non-High Density Lipoprotein (HDL) cholesterols | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of non-HDL cholesterol.
CagriSema versus semaglutide: CGM - Change in Time In Range (TIR) 3.9-10.0 mmol/L (70-180 mg/dL) | From baseline (week -3) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: Ratio to baseline in high sensitivity C-Reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of hsCRP.
CagriSema versus semaglutide: Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 68)
  Measured in mmol/L.
CagriSema versus semaglutide: Achievement of HbA1c target values of less than (<) 7.0% (<53 millimoles per mole [mmol/mol]) | At end of treatment (week 68)
  Measured as count of participants.
CagriSema versus semaglutide: Achievement of HbA1c target values of less than or equal to (≤)6.5% (≤48 mmol/mol) | At end of treatment (week 68)
  Measured as count of participants.
CagriSema versus semaglutide: CGM - Change in time above range, >10.0 mmol/L (>180 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: CGM - Change in time above range, >13.9 mmol/L (>250 mg/dL) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage-points.
CagriSema versus semaglutide: CGM - Within-day glycaemic variability (% coefficient of variation [CV]) | At end of treatment (week 68)
  Measured in percentage.
CagriSema versus semaglutide: Achievement of ≥ 5 % weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants.
CagriSema versus semaglutide: Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimetre.
CagriSema versus semaglutide: Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in mmHg.
CagriSema versus semaglutide: Ratio to baseline in total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of total cholesterol.
CagriSema versus semaglutide: Ratio to baseline in HDL cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of HDL cholesterol.
CagriSema versus semaglutide: Ratio to baseline in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of LDL cholesterol.
CagriSema versus semaglutide: Ratio to baseline in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of VLDL.
CagriSema versus semaglutide: Ratio to baseline in free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Measured as ratio of free fatty acids.
CagriSema versus semaglutide: Change in Short Form (SF)-36v score- Physical component summary score | From baseline (week 0) to end of treatment (week 68)
  SF-36v2 measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and an standard deviation of 10. Physical component summary score range from 6.1 to 79.7, with higher scores indicating better functional health and well-being.
CagriSema versus semaglutide: Change in SF-36v2 score- Mental component summary score | From baseline (week 0) to end of treatment (week 68)
  SF-36v2 measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and an standard deviation of 10. Mental component summary score range from -3.8 to 78.7, with higher scores indicating better functional health and well-being.
CagriSema versus semaglutide: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score | From baseline (week 0) to end of treatment (week 68)
  DTSQc measures treatment satisfaction and diabetes-specific quality of life (QoL). The measure consists of 8 items yielding 1 global score and 2 single item scores. Total treatment satisfaction scores range from 0-36, with higher scores indicating greater satisfaction; the perceived frequency of hyperglycemia/hypoglycemia items are scored separately, with lower scores indicating better perceived blood glucose control.
CagriSema versus semaglutide: Change in Treatment Related Impact Measure for Diabetes (TRIM-D) score | From baseline (week 0) to end of treatment (week 68)
  TRIM-D measures impact of diabetes treatment. The measure consists of 28 items yielding 5 domain scores and a total score. The scores were transformed to a 0-100 scale with higher scores indicating a better health state.
CagriSema versus semaglutide, placebo and cagrilintide: Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 75)
  Measured as count of events.
CagriSema versus semaglutide: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline (week 0) to end of study (week 75)
  Measured as count of episodes.
CagriSema versus semaglutide: Number of severe hypoglycaemic episodes (level 3) | From baseline (week 0) to end of study (week 75)
  Measured as count of episodes. Hypoglycaemia episodes (level 3) are the episodes associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (403):
- United States (100):
  - Synexus Clin Res-Birmingham, Birmingham, Alabama
  - Univ of Alabama_Birmingham, Birmingham, Alabama
  - Cahaba Research, Pelham, Alabama
  - Velocity Clinical Research-Phoenix, Phoenix, Arizona
  - Synexus Rsch /Cnt Phnx Med C, Phoenix, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Res-Banning, Banning, California
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - John Muir Physicians Network, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Velocity Clin Res Gardena, Gardena, California
  - Velocity Clin Res San Diego, La Mesa, California
  - Loma Linda Univ Hlth Cr Endo, Loma Linda, California
  - Facey Medical Foundation, Mission Hills, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Velocity Clin Res- San Bern, San Bernardino, California
  - Linda Vista Health Care Ctr, San Diego, California
  - Velocity Clin Res Santa Ana, Santa Ana, California
  - Premier Medical Center, Inc., Toluca Lake, California
  - Velocity Clin Res - Panorama, Van Nuys, California
  - Optumcare Clinical Trials,LLC-Golden, Colorado Springs, Colorado
  - Northeast Research Institute, Jacksonville, Florida
  - Clinical Trial Services Corp, Miami, Florida
  - Bioclinical Research Alliance, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - South Broward Research LLC, Miramar, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Optimal Research Sites, Orange City, Florida
  - Advent Health-Res Inst, Orlando, Florida
  - AdventHealth Diab Inst, Orlando, Florida
  - Synexus Clin Res - Orlando, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - East Coast Institute for Res, Macon, Georgia
  - Urban Family Practice Assoc, Marietta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Pacific Diabetes & Endo Ctr, Honolulu, Hawaii
  - St. Luke's Health System, Boise, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Endeavor Health, Skokie, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Iowa Diabetes & Endo Res Ctr, West Des Moines, Iowa
  - Alliance for Multispec Res, Newton, Kansas
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - Velocity Clin Res Lafayette, Lafayette, Louisiana
  - BTC of New Bedford, LLC, New Bedford, Massachusetts
  - Velocity Clin Res Gulfport, Gulfport, Mississippi
  - Diabetes & Endo Specialists Inc, Chesterfield, Missouri
  - Premier Research Inc., Trenton, New Jersey
  - Velocity Clin Res Albuquerque, Albuquerque, New Mexico
  - AMC Community Endocrinology, Albany, New York
  - Velocity Clin Res Syracuse, East Syracuse, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Radiant Research Inc. - Akron, Akron, Ohio
  - Centricity Research, Columbus, Ohio
  - Alliance for Multispec Res, Norman, Oklahoma
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Velocity Clin Res Providence, East Greenwich, Rhode Island
  - AnMed Health IMA, Anderson, South Carolina
  - Synexus Clin Res US-Anderson, Anderson, South Carolina
  - Velocity Clinical Res-Anderson, Anderson, South Carolina
  - Velocity Clin Res Gaffney, Gaffney, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Velocity Clin Res Spartanburg, Spartanburg, South Carolina
  - Holston Medical Group Pc, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Velocity Clin Res Austin, Austin, Texas
  - UT Health University of Texas, Bellaire, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Synexus Clin Res Dallas, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - JCCT- Juno NW Houston, Houston, Texas
  - Synergy Groups Medical, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Medical Colleagues-Texas LLP, Katy, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Discovery MMS Services, INC, Missouri City, Texas
  - AES San Antonio, San Antonio, Texas
  - University of Texas San Antonio, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - DM Clin Rsrch/Fam Diag Clinic, Tomball, Texas
  - Diabetes & Endo Treatment Spec, Sandy City, Utah
  - Velocity Clin Res-Salt Lk City, West Jordan, Utah
  - TPMG Clinical Research, Newport News, Virginia
  - Rainier Clin Res Ctr Inc, Renton, Washington
  - St. Vincent Hosp-Prevea Health, Green Bay, Wisconsin
- Argentina (6):
  - Mautalen Salud e investigación, CABA, Buenos Aires
  - Sanatorio Güemes, CABA, City of Buenos Aires
  - Instituto de Investigaciones Clínicas Rosario, Rosario, Santa Fe Province
  - STAT Research, Buenos Aires
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, CABA
- Australia (8):
  - Charles Perkins Centre, Camperdown, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Logan Hospital, Meadowbrook, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - St Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
- Brazil (3):
  - Cline Research Center, Curitiba, Paraná
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
- Bulgaria (10):
  - IPSMC - Dr. Nikolay Kostadinov EOOD, Burgas
  - Dr. Tatyana Metalova - AIPSMCE EOOD, Gotse Delchev
  - ASOMCEID - Individual Practice - Dr. Abdul-Azis EOOD, Kardzhali
  - Medical Center Zdrave Lom EOOD, Lom
  - Medical Centre Razgrad OOD, Razgrad
  - DCC Ascendent OOD, Sofia
  - Medical Center Maraya Med EOOD, Sofia
  - Medical Centre - Clinic Nova EOOD, Varna
  - Medical centre Clinic Nova, Varna
  - UMHAT Sveta Marina EAD, Varna
- Canada (31):
  - Centricity Research Calgary Endocrinology, Calgary, Alberta
  - Centricity Research Calgary, Calgary, Alberta
  - Synergy Wellness Clinic, Sherwood Park, Alberta
  - Guilford Med Clinic, Surrey, British Columbia
  - TLC Diabetes and Endocrinology, Surrey, British Columbia
  - Ocean West Research Clinic, Surrey, British Columbia
  - Hilltop Medical Clinic, Surrey, British Columbia
  - Spectrum Health Clinic, Vancouver, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Centricity Res. Barrie Endo, Barrie, Ontario
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Centricity Research Vaughn Endocrinology, Concord, Ontario
  - Medical Trust Clinics, Inc., Courtice, Ontario
  - Centricity Research Etobicoke Endocrinology, Etobicoke, Ontario
  - Milestone Research, London, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - My Endo Diabetes & Endo Cent, Markham, Ontario
  - Centricity Research Ottawa LMC, Nepean, Ontario
  - Centricity Research Oshawa, Oshawa, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Centre Medical Acadie, Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
  - Q & T Research Sherbrooke Inc., Sherbrooke, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Diex Recherche Quebec Inc., Québec
  - Clin des Mal Lipid de Quebec, Québec
  - Centre de Recherche Saint-Louis, Québec
- China (9):
  - Beijing Friendship Hospital, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Huaihe Hospital of Henan University-Endocrinology, Kaifeng, Henan
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - Suzhou Municipal Hospital-Endocrinology, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'Nan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
- Colombia (4):
  - FOSCAL, Floridablanca, Santander Department
  - Cimedical, Barranquilla
  - Clinica Imbanco SAS, Cali
  - IMAT - Oncomedica, Montería
- Croatia (6):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Poliklinika SLAVONIJA OSIJEK, Osijek, County of Osijek-Baranja
  - Clinical Hospital Centre Rijeka_Endocrinology, Rijeka, Primorje-Gorski Kotar County
  - Specijalna bolnica Thalassotherapia, Opatija
  - General Hospital Dr. Josip Bencevic_Diabetic department, Slavonski Brod
  - Opca bolnica Varazdin_Endocrinology, Varaždin
- Czechia (7):
  - IKEM Centrum Diabetologie, Prague, Czech Republic
  - Fakultní nemocnice U sv. Anny v Brně, Brno
  - Edumed Broumov, Broumov
  - Diahaza s.r.o., Holešov
  - DIALINE s.r.o., Plzeň 3
  - Diabet2 s.r.o., Prague
  - MUDr. Michala Pelikanova, Prague
- Denmark (6):
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus N
  - Bispebjerg Hospital, IC-Forskning, Copenhagen
  - Steno Diabetes Center Copenhagen, Herlev
  - Hillerød Endokrinologisk amb. H0652, Hillerød
  - Hvidovre Hospital Endokrinologisk forsk. afs. 159, Hvidovre
  - Steno Diabetes Center Odense, Odense C
- Finland (5):
  - Terveystalo Jyväskylä, Jyväskylä
  - Seinäjoen keskussairaala, Seinäjoki
  - Pihlajalinna Koskiklinikka, Tampere
  - Terveystalo Tampere Rautatienkatu, Tampere
  - Turku University Hospital, Turku
- Germany (15):
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - Diabetologische Schwerpunktpraxis Daaden, Daaden
  - Diabeteszentrum-Do Dres. K U. Ch. Busch GbR, Dortmund
  - Uniklinik TU Dresden - Med. Klinik III, Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - MVZ Diabeteszentrum Dr. Tews GmbH, Gelnhausen
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Diabetes Zentrum Wandsbek Berufsausuebungsgemeinschaft GbR, Hamburg
  - Diabetologische Gemeinschaftspraxis Dr. Staudenmeyer und Dr. Schiwietz, Lingen
  - Die Praxis am Ludwigsplatz, Ludwigshafen
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Medicover Neuroendokrinologie MVZ München, München
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis für Innere Medizin - Zwenkau, Zwenkau
- Greece (10):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - General Hospital Of Thessaloniki Papageorgiou, Nea Efkarpia, Thessaloniki
  - Iatriko Psychicou Private Clinic, Athens
  - "Laiko" General Hospital of Athens, Athens
  - General hospital of Athens 'G.Gennimatas', Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Univ Gen Hospital Larisa, Larissa
  - "AHEPA" University Hospital of Thessaloniki, Thessaloniki
  - NextHealth S.A. - Department of Endocrinology, Metabolism & Diabetes, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
- Hungary (9):
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged, Csongrád-Csanád
  - Debreceni Egyetem Belgyógyászati Klinika, Debrecen, Hajdú-Bihar
  - Óbudai Egészségügyi Centrum, Budapest, Pest County
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MH Egészségügyi Központ, Budapest
  - Kaposi Mór Oktató Kórház, Kaposvár
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Vas Vármegyei Markusovszky Egyetemi Oktatókórház, Szombathely
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- India (15):
  - Yalamanchi Hospitals and Research centres pvt ltd, Vijaywada, Andhra Pradesh
  - Gauhati Medical College and Hospital, Guwahati, Assam
  - Swasthya Diabetes Care, Ahmedabad, Gujarat
  - Lifecare Hospital and Research Centre, Bengaluru, Karnataka
  - K R Hospital, Mysuru, Karnataka
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Ashirwad Hospital and Research Centre, Thane, Maharashtra
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - KG Hospital, Coimbatore, Tamil Nadu
  - Gleneagles Hospitals, Hyderabad, Telangana
  - Dr P V Rao - Diabetes Research Centre, Hyderabad, Telangana
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education & Research, Chandigarh
  - Lady Hardinge Medical College, New Delhi
- Israel (9):
  - Clalit sick fund Herzeliya, Herzeliya, Israel
  - Linn clinic - Clalit Health Services, Haifa
  - Linn clinic - Diabetes Unit, Haifa
  - Clalit sick fund Herzlia, Herzliya
  - Wolfson MC - Diabetes Clinic, Holon
  - Hadassah Ein Karam MC - Diabetes Unit, Jerusalem
  - Kaplan MC - Metabolic Unit, Rehovot
  - Kaplan MC, Rehovot
  - Sheba MC - Endocrinology Clinic, Tel Litwinsky
- Italy (14):
  - AOU Careggi Firenze, Florence, Fi
  - Istituto Scientifico San Raffaele, Milan, MI
  - AOU Careggi Firenze, Florence, Tuscany
  - Azienda Sanitaria Usl Toscana Sud Est - Ospedale San Donato, Arezzo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti Scalo
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - AOUP Giaccone Palermo, Palermo
  - Dip. di Medicina Interna Policlinico Universitario Palermo, Palermo
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di scienze Mediche e Chirurgiche, Rome
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Civile Maggiore Borgo Trento, Verona
- Japan (10):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Fukushima, Japan
  - Abe Diabetes Clinic_Internal Medicine, Ōita, Oita, Japan
  - Akaicho Clinic, Chiba-shi, Chiba
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - Minami Akatsuka Clinic, Mito-shi, Ibaraki
  - Medical Research Institute KITANO HOSPITAL_Diabetes & Endocrinology, Osaka-shi, Osaka
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
- Mexico (4):
  - Centro de investigación en Artritis y Osteoporosis S.C., Mexicali, Estado de Baja California
  - InstitutoJalisciense de Investigación en Diabetes y Obesidad, Guadalajara, Jalisco
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - Centro de Estudios de Investigación Metabólicos y Cardio, Ciudad Madero, Tamaulipas
- Poland (20):
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów, Masovian Voivodeship
  - Instytut Diabetologii Sp. z o.o., Warsaw, Mazovian Voivodeship
  - Centrum Medyczne Medyk Sp. z o.o., Rzeszów, Podkarpackie Voivodeship
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - PAKS III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Dąbrowa Górnicza, Silesian Voivodeship
  - PAKS III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Tychy, Silesian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - PAKS III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Dąbrowa Górnicza
  - Velocity Nova Sp. z o.o., Lublin
  - KO-MED Centra Kliniczne Sp. z o.o., Puławy
  - Velocity Nova Sp. z o.o., Staszów
  - NBR Polska Tomasz Klodawski, Warsaw
  - Instytut Diabetologii Sp. z o.o., Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Zgierskie Centrum Kardiologii Med-Pro Polsko-Amerykańskich Klinik Serca, Zgierz
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Lodz, Łódź Voivodeship
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Romania (15):
  - Cabinet Medical Individual Dr. Ramona Dragut SRL, Piteşti, Argeş
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Spitalul Clinic Judetean Urgenta Cluj-Napoca, Cluj-Napoca, Cluj
  - Poli Cardinal Med Srl, Reghin, Mureș County
  - Diabmed Dr Popescu Alexandrina SRL, Ploieşti, Prahova
  - CMI Dr. Busegeanu Mihaela Magdalena, Ploieşti, Prahova
  - Cabinet Medical de Diabet, Nutritie si Boli Metabolice-Dr. Zaharie Daniela Gabriela, Zalău, Sălaj County
  - CMI Dr. Pletea Noemi SRL, Bacau
  - Mariodiab Clinic SRL, Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - Diabet Med SRL, Bucharest
  - Urodiamed SRL, Craiova
  - S.C Milena Sante SRL, Galati
  - Gama Diamed Srl, Mangalia
  - Bella Praxis S.R.L., Paşcani
- Serbia (6):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocr, Kragujevac
- Slovakia (11):
  - DIADA, s.r.o., Bardejov
  - Diabetologicka ambulancia DIOLI s.r.o., Košice
  - DIOLI s.r.o., Košice
  - MediVet s.r.o., Malacky
  - DIALIPID, s.r.o., Prešov
  - MUDr. Jan Culak, s.r.o., Prievidza
  - DIACENTRUM, s.r.o., Ružomberok
  - MEDI-DIA s.r.o., Sabinov
  - DEImedi, s. r. o., Šurany
  - ARETEUS s.r.o., Trebišov
  - iDia s. r. o., Žiar nad Hronom
- Slovenia (8):
  - Healthcare centre Kocevje, Kočevje
  - Healthcare Centre Koper, Koper
  - Dermatologija Bartenjev, Ljubljana
  - UKC Ljubljana, Endocrinology and Diabetes, Ljubljana
  - UKC Maribor - diabetes, Maribor
  - Healthcare Centre Nova Gorica, Nova Gorica
  - General Hospital Nova Gorica_Diabetes, Šempeter pri Gorici
  - Hospital Topolšica, Topolšica
- South Africa (6):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Sandton Medical Research, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Paarl Research Centre, Paarl, Cape Town, Western Cape
- South Korea (7):
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Yeungnam University Medical Center, Daegu
  - Chosun University Hospital, Gwangju
  - Kyunghee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - ABS La Roca del Vallés_Endocrinología, La Roca Del Vallés
  - Hospital Universitario de Móstoles, Móstoles
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital General de Segovia, Segovia
  - Hospital Infanta Luisa, Seville
  - Hospital La Fe - Endocrinología y Nutrición, Valencia
- Sweden (7):
  - CTC EbbePark Linköping, Linköping
  - Clemenstorgets Hjärtmottagning, Lund
  - Endokrinologkliniken, Lund, Lund
  - Forskningsmottagning Internmedicin (tidigare KFE), Malmo
  - CTC GoCo Mölndal, Mölndal
  - Örebro UH - Överviktsenheten, Örebro
  - Karolinska Universitetssjukhuset Solna,FOU Tema Hjärta Kärl, Stockholm
- Taiwan (2):
  - Changhua Christian Hospital_Metabolic Dept., Changhua
  - Taipei Medical University Hospital, Taipei
- Turkey (Türkiye) (20):
  - Cukurova Universitesi Tip Fakultesi, Adana
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Endokrinoloji, Adana
  - Akdeniz University Tip Fakultesi Hastanesi, Antalya
  - Akdeniz Üniversitesi Hastanesi- Endokrinoloji, Antalya
  - Eskisehir Osmangazi University School of Medicine, Eskişehir
  - Eskişehir Osmangazi Üniversitesi Sağlık, Uygulama ve Araştırma Hastanesi, Eskişehir
  - Haseki Eğitim ve Araştırma Hastanesi- Dahiliye, Istanbul
  - Haseki Sultangazi, Istanbul
  - Seyrantepe Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi- Seyrantepe Yerleşkesi- Endokrinoloji, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi - Endokrinoloji, Istanbul
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Endokrinoloji, Istanbul
  - Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul
  - Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - T.C SB Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Recep Tayyip Erdoğan Üni. Eğitim ve Araştırma Hastanesi, Rize
  - Recep Tayyip Erdoğan Üniversitesi EAH-Endokrinoloji, Rize
  - Tekirdag Namık Kemal UTF, Tekirdağ
  - Tekirdağ Namık Kemal Üniversitesi Hastanesi- Dahiliye, Tekirdağ
- United Kingdom (12):
  - Lister Hospital, Stevenage, Hertfordshire
  - Pickering Medical Practice, Pickering, North Yorkshire
  - Aberdeen Royal Infirmary - Diabetes, Aberdeen
  - Aberdeen Royal Infirmary, Aberdeen
  - Oldfield Surgery, Bath
  - Oakenhurst Medical Practice, Blackburn
  - Ninewells Hospital, Dundee
  - Aintree University Hospital, Liverpool
  - Norfolk and Norwich University Hospital Trust, Norwich
  - Moorgreen Hospital, Southampton
  - Joint Clinical Research Facility - Swansea, Swansea
  - Royal Cornwall Hospital (Treliske), Truro

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com